CLINICAL TRIAL: NCT02971839
Title: A Phase 2, Randomized, Parallel-Group, Double-Blind, Placebo Controlled Study to Evaluate the Safety and Efficacy of CTP-656 With an Open-Label Active Comparator in Patients With Cystic Fibrosis With CFTR Gating Mutations.
Brief Title: Study to Evaluate the Safety and Efficacy of CTP-656 in Patients With Cystic Fibrosis With CFTR Gating Mutations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision by Sponsor.
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP656.2001
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Results first posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- VX-561 20 mg (Experimental)
  Interventions: Drug: VX-561
- VX-561 100 mg (Experimental)
  Interventions: Drug: VX-561
- VX-561 150 mg (Experimental)
  Interventions: Drug: VX-561
- Ivacaftor (Active Comparator)
  Interventions: Drug: IVA
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VX-561
  Other Names: CTP-656
  Arms: VX-561 100 mg; VX-561 150 mg; VX-561 20 mg
Drug: Placebo
  Arms: Placebo
Drug: IVA
  Other Names: ivacaftor; VX-770; Kalydeco
  Arms: Ivacaftor

SUMMARY:
This study will evaluate the efficacy and safety of CTP-656 in patients with cystic fibrosis (CF) who have a cystic fibrosis transmembrane conductance regulator (CFTR) gating mutation.

DETAILED DESCRIPTION:
This is a randomized, parallel-group, double-blind, placebo controlled multicenter study to evaluate the safety and efficacy of CTP-656 in CF patients with CFTR gating mutations, compared to Kalydeco, for a total of 28 days. Subjects will be randomized to receive either double-blind CTP-656 or placebo, or open-label Kalydeco.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Has a confirmed diagnosis of CF with at least one allele of the following CFTR gating mutations: G551D, G1244E, G1349D, G178R, G551S, S1251N, S1255P, S549N, and S549R.
* Has been stable on Kalydeco therapy for at least 3 months prior to screening
* Has FEV1 ≥ 60% of predicted normal for age, sex, and height at screening and baseline (Day 1) assessments
* Weighs at least 40 kg at screening
* Patients of either gender and women of childbearing potential must be willing to use a medically highly effective form of birth control during the treatment period and 30 days after the last dose of study treatment.

Exclusion Criteria:

* Acute upper respiratory infection or lower respiratory infection, pulmonary exacerbation, or changes in therapy within 4 weeks of study treatment
* Uncontrolled type 2 diabetes, or uncontrolled CF-related diabetes
* History of hepatitis C or chronic active hepatitis B infection
* History of pulmonary tuberculosis, non-tuberculosis mycobacterial infections or allergic bronchopulmonary aspergillosis (ABPA) treated during screening or within 2 years prior to screening
* Colonization with B. cenocepacia, B. dolosa, B. multivorans, and/or M. abcessus within 2 years prior to Screening
* Abnormal liver function
* History of abnormal renal function
* History of prolonged QTcF > 450 msec for males or QTcF > 470 msec for females
* History of solid organ or hematological transplantation
* Using any inhibitor or inducer of cytochrome P450/3A during the study or within 30 days of screening
* Women who are pregnant or lactating, or have plans to become pregnant during the study or within 1 month following the last dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - University of Southern California, Los Angeles, California
  - Stanford Hospital, Palo Alto, California
  - Children's National Health, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Rush University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Washington University, St Louis, Missouri
  - Atlantic Health, Morristown, New Jersey
  - New York Medical College, Valhalla, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- VX-561 20 mg: Participants received VX-561 20 mg orally once daily for 28 days.
- VX-561 100 mg: Participants received VX-561 100 mg orally once daily for 28 days.
- VX-561 150 mg: Participants received VX-561 150 mg orally once daily for 28 days.
- Placebo: Participants received placebo matched to VX-561 orally once daily for 28 days.
- Ivacaftor: Participants received Ivacaftor 150 mg orally every 12 hours for 28 days.
Period: Overall Study
Arm/Group | VX-561 20 mg | VX-561 100 mg | VX-561 150 mg | Placebo | Ivacaftor
Started | 2 | 2 | 2 | 2 | 3
Completed | 2 | 2 | 2 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VX-561 20 mg | VX-561 100 mg | VX-561 150 mg | Placebo | Ivacaftor | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.0 (1.41) | 20.0 (1.41) | 19.5 (2.12) | 29.0 (2.83) | 19.7 (0.58) | 22.2 (4.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 2 | 2 | 9
  Male | 0 | 1 | 0 | 0 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 2 | 2 | 1 | 3 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 2 | 2 | 2 | 3 | 11
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Sweat Chloride [Mean (Standard Deviation); unit: millimole per liter (mmol/L)] | 59.25 (16.617) | 82.25 (27.931) | 61.50 (32.527) | 36.50 (29.698) | 71.25 (37.830) | 62.15 (27.355)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Sweat Chloride at Day 28
Time Frame: From baseline at Day 28
Population: As pre-specified in SAP section 4.13 (Changes in Conduct or Planned Analyses), due to the limited number of participants being enrolled in the study, model-based analyses and summary statistics plan were not performed. Therefore, no efficacy summary is provided for this outcome measure.
Arm/Group | VX-561 20 mg | VX-561 100 mg | VX-561 150 mg | Placebo | Ivacaftor
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) at Day 28
Time Frame: From baseline at Day 28
Population: As pre-specified in SAP section 4.13 (Changes in Conduct or Planned Analyses), due to the limited number of participants being enrolled in the study, all model-based analyses and summary statistics are no longer applicable and are therefore removed from analysis plan. Therefore no efficacy summary is available for this outcome measure.
Arm/Group | VX-561 20 mg | VX-561 100 mg | VX-561 150 mg | Placebo | Ivacaftor
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in Cystic Fibrosis Questionnaire-Respiratory Domain (CFQ-R) at Day 28
Time Frame: From baseline at Day 28
Population: as for outcome 2
Arm/Group | VX-561 20 mg | VX-561 100 mg | VX-561 150 mg | Placebo | Ivacaftor
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 35
Arm/Group | VX-561 20 mg | VX-561 100 mg | VX-561 150 mg | Placebo | Ivacaftor
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 1/2 | 2/2 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VX-561 20 mg (N=2) | VX-561 100 mg (N=2) | VX-561 150 mg (N=2) | Placebo (N=2) | Ivacaftor (N=3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Forced expiratory volume decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 1 | 0
Pulmonary function test decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-10-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT02971839/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT02971839/SAP_001.pdf